CLINICAL TRIAL: NCT02326012
Title: Emotion Regulation Individual Therapy for Adolescents With NSSI - An Open Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1-31/3
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Nonsuicidal Self-Injury
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emotion Regulation Individual Therapy for Adolescents (Experimental)
  Interventions: Behavioral: Emotion Regulation Individual Therapy for Adolescents

INTERVENTIONS:
Behavioral: Emotion Regulation Individual Therapy for Adolescents

SUMMARY:
The primary aim is to investigate the effectiveness of Emotion Regulation Individual Therapy for Adolescents (ERITA) who self-harm.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of NSSI as defined by DSM-5 Section 3
* < 1 NSSI episode during the past month
* at least one parent needs to commit to participate in the parent program

Exclusion Criteria:

* bipolar disorder I or primary psychosis
* severe suicidal ideation
* ongoing substance dependence
* Insertion/withdrawal of psychopharmacological substances within two months prior to the treatment
* other acute primary axis I diagnosis (e.g. anorexia nervosa) that demand treatment in first hand
* current life circumstances that would hinder the treatment (i.e. ongoing domestic abuse)
* insufficient Swedish language skills
* Cocurrent treatment with Mentalization based therapy (MBT) or Dialectical behavioral therapy (DBT)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Deliberate Self-Harm Inventory - 9 item version | Baseline (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in self-harming behaviors when measures weekly, after 12 weeks and at 6 months after treatment has ended.

SECONDARY OUTCOMES:
Borderline Symptom List Behavior supplement (BSL-supplement) | Baseline (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in self-destructive and risky behaviors when measures weekly, after 12 weeks and at 6 months after treatment has ended.
Difficulties in Emotion Regulation Scale -16 item version (DERS-16) | Baseline (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in difficulties in emotion regulation when measures weekly, after 12 weeks and at 6 months after treatment has ended.
Diary questionnaire (DQ) | Baseline (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in difficulties in emotion regulation when measures weekly, after 12 weeks and at 6 months after treatment has ended.
Difficulties in Emotion Regulation Scale (DERS) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in difficulties in emotion regulation after 12 weeks and at 6 months after treatment has ended.
Strengths and Difficulties Questionnaire Child and Parent version (SDQ-C/P) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in strengths and difficulties after 12 weeks and at 6 months after treatment has ended.
Borderline personality features in childhood (BPFS-C) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in borderline personality features after 12 weeks and at 6 months after treatment has ended.
The alcohol use disorders identification test - C (AUDIT-C) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in alcohol use after 12 weeks and at 6 months after treatment has ended.
Evaluation of the Drug Use Disorders Identification Test - C (DUDIT-C) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from baseline in drug use after 12 weeks and at 6 months after treatment has ended.

OTHER OUTCOMES:
Euroqol-5D (EQ-5D) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from Baseline in quality of life after 14 weeks and at 6- and 12 months after treatment has Change from baseline in quality of life after 12 weeks and at 6 months after treatment has ended. Used for health economic evaluations.
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness - Child version (TiC-P) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change from Baseline in societal costs after 14 weeks and at 6- and 12 months after treatment has Change from baseline in quality of life after 12 weeks and at 6 months after treatment has ended. Used for health economic evaluations.
Patient Health Questionnaire (PHQ9) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change in patient parent health from baseline after 12 weeks and at 6 months after treatment has ended.
General Anxiety Disorder (GAD7) | Baseline (7 days prior to treatment start), post-treatment (12 weeks) and six months follow-up
  Change in patient parent health from baseline after 12 weeks and at 6 months after treatment has ended.
The treatment credibility scale | One week after treatment start
  Perceived treatment credibility
Working Alliance Inventory (WAI) short version | Three weeks after treatment start
  Perceived working alliance

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Bjureberg J, Sahlin H, Hellner C, Hedman-Lagerlof E, Gratz KL, Bjarehed J, Jokinen J, Tull MT, Ljotsson B. Emotion regulation individual therapy for adolescents with nonsuicidal self-injury disorder: a feasibility study. BMC Psychiatry. 2017 Dec 28;17(1):411. doi: 10.1186/s12888-017-1527-4. PMID 29282024